CLINICAL TRIAL: NCT00395551
Title: A Single Center Study of the Safety and Efficacy of Multiple Intravitreal Injections of Ranibizumab in Subjects With CNV Secondary to Causes Other Than AMD.
Brief Title: Safety Study of Ranibizumab Eye Injections to Treat Choroidal Neovascularization That Was Caused Other Than by Age-Related Macular Degeneration.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ophthalmic Consultants of Boston (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Dr. Jeffrey S. Heier, Ophthalmic Consultants of Boston
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FVF 3688 Non-AMD
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Choroidal Neovascularization
Keywords: choroidal neovascularization; Choroidal Neovascularization Not related to Age-Related Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ranibizumab (Active Comparator): ranibizumab 0.5mg intravitreal injection
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg intravitreal injection

SUMMARY:
The purpose of this study is to determine whether ranibizumab is effective in the treatment of choroidal neovascularization secondary to causes other then wet macular-degeneration.

ELIGIBILITY:
Inclusion Criteria:

* active choroidal neovascularization

Exclusion Criteria:

* pregnancy,age-related macular degeneration, current eye infection or recent eye surgery, participating in other eye studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures for safety and tolerability | Mean change in visual acuity from baseline to 6 months & 12 months

SECONDARY OUTCOMES:
The secondary outcome measures for efficacy | Mean change in visual acuity from baseline to 6 & 12 months. Change in retinal thickness from baseline to week 1, month 1, 2, 3, 6, & 12 measured by OCT. Change in area of CNV from baseline to month 3, 6 & 12 measured by FA

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, M.D., Principal Investigator — Ophthalmic Consultants of Boston